CLINICAL TRIAL: NCT06285604
Title: Effect Evaluation of Different Blood Products Infusion on Neonatal Anemia
Status: Active, not recruiting | Type: Observational
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Principal Investigator, Guangyong Ye, Doctor, Women's Hospital School Of Medicine Zhejiang University
Other Study IDs: IRB-20230398-R
Record Dates: First submitted 2024-01-28; First posted 2024-02-29 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-02

CONDITIONS: Neonatal Anemia
MeSH Terms: conditions — Anemia, Neonatal | interventions — Blood Transfusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- IRBC: Anemic neonates with irradiated red blood cells transfusions.
  Interventions: Procedure: Blood transfusion
- WRBC: Anemic neonates with washed red blood cells transfusions.
  Interventions: Procedure: Blood transfusion
- LPRBC: Anemic neonates with leukocyte privative red blood cells transfusions.
  Interventions: Procedure: Blood transfusion

INTERVENTIONS:
Procedure: Blood transfusion — Transfusion of designated red blood cell products to anemic neonates.

SUMMARY:
The goal of this observational study is to evaluate the clinical efficacy of the transfusion of irradiated red blood cells, washed red blood cells, and leukocyte privative red blood cells, and to study the changes of inflammatory response before and after the transfusion of irradiated red blood cells, washed red blood cells, and leukocyte privative red blood cells in anemic neonates. The main questions it aims to answer are:

* Objective evaluation of the advantages and disadvantages of transfusion of different blood products in the treatment of neonatal anemia from the clinical efficacy.
* To provide objective basis for clinical rational use of blood in the selection of blood products.

Participants will be transfused with fresh irradiated red blood cells, washed red blood cells, and leukocyte privative red blood cells respectively according to relevant clinical and laboratory indicators.

ELIGIBILITY:
Inclusion Criteria:

Neonates with stable hemodynamics who need blood transfusion are comprehensively evaluated by neonatologists according to their clinical conditions (heart, respiratory status, postnatal age, pregnancy at birth), laboratory indicators, etc. Diagnosis of Neonatal Septicemia:

* The mother had chorioamnionitis infection or Premature rupture of membranes (PROM) ≥18 h.
* The clinical diagnosis is that there are clinical abnormal manifestations, and any of the following conditions is met at the same time: ① blood non-specific examination ≥ 2 items are positive, ② cerebrospinal fluid examination is purulent meningitis change, and ③ pathogenic bacteria DNA is detected in blood.
* The diagnosis was confirmed as having clinical manifestations and positive blood culture or cerebrospinal fluid (or other sterile cavity fluid) culture.

Exclusion Criteria:

* Infants with necrotizing enterocolitis (NEC) (current or previous).
* Feeding intolerance (defined as the decision of the treatment clinical team to suspend feeding / suspend feeding for at least 12 hours).
* RBC transfusion in the past 72 hours; Children who received ibuprofen / indomethacin / surgery 72 hours ago and / or severe congenital malformations such as congenital gastrointestinal tract, complex cardiopulmonary / fatal abnormalities or need emergency blood transfusion.

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates who received blood transfusion at the Women's Hospital School of Medicine Zhejiang University from October 1, 2023 to September 30, 2025.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy of different red blood cell products transfusion in anemic neonates | The test results of each subject before and 24 hours after blood transfusion were analyzed.
  The changes of hemoglobin concentration, crSo2 and cFTOE before and after transfusion were detected to evaluate the effects of different red blood cell products on brain oxygenation capacity of anemic neonates.
The changes of inflammatory response before and after transfusion in anemic neonates | The test results of each subject before and 24 hours after blood transfusion were analyzed.
  IL-6, IL-10 and CRP levels were measured, and the effect of infusion of different red blood cell products on the potential inflammatory response of anemic neonates was evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No